CLINICAL TRIAL: NCT04844086
Title: Infusion of CD19-Specific Chimeric Antigen Receptor T-cells Produced by Rapid Personalized Manufacture for Patients With Advanced Lymphoid Malignancies
Brief Title: RPM CD19-mbIL15-CAR-T Cells in Patient With Advanced Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: CAR-T manufacturing technology can not meet the dose requirement for clinical patients.
Sponsor: Eden BioCell Ltd. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eden 2020-01
Record Dates: First submitted 2021-04-06; First posted 2021-04-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma, Relapsed; Non-Hodgkin's Lymphoma Refractory; Primary Mediastinal Large B Cell Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; High-grade B-cell Lymphoma
Keywords: CD19 specific CAR; Autologous
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Recurrence; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infusion RPM CD19-mbIL15-CAR-T cell (Experimental): In this study, anti-CD19 autologous chimeric antigen receptor T-cells infusion produced by rapid personalized manufacture are used to treat patients with relapsed/refractory Advanced Lymphoid Malignancies.
  Route of administration: Intravenous injection.
  Lymphodepletion conditioning:
  Lymphodepletion will be conducted several days prior to RPM CD19-mbIL15-CAR-T cell infusion.
  A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  Interventions: Biological: RPM CD19-mbIL15-CAR-T cells

INTERVENTIONS:
Biological: RPM CD19-mbIL15-CAR-T cells — Single dose of RPM CD19-mbIL15-CAR-T cells will be infused, and a standard "3+3" design will be applied.
  Drug: Fludarabine
  Fludarabine is used for lymphodepletion.
  Drug: Cyclophosphamide
  Cyclophosphamide is used for lymphodepletion

SUMMARY:
This is an open-label Phase 1 study to determine the feasibility, safety, and the recommended maximum tolerated Dose (MTD) of a single infusion of RPM CD19 mbIL15 CAR-T cells for adult patients. Approximately 24 subjects will be enrolled and it is anticipated approximately 16 subjects will be infused at the varied doses of T cells.

DETAILED DESCRIPTION:
This is an open-label Phase 1 study to determine the feasibility, safety, and the recommended maximum tolerated Dose (MTD) of a single infusion of RPM CD19 mbIL15 CAR-T cells for adult patients. Approximately 24 subjects will be enrolled and it is anticipated approximately 16 subjects will be infused at the varied doses of T cells.

This study will very rapidly administer T cells that are genetically modified by electroporation using DNA plasmids from the SB system to co-express CD19RCD8CD28 (the CAR), mbIL15, and HER1t. The presence of mbIL15 may allow for reduced doses of CAR-T cells to be infused to reduce the risk for adverse events, such as cytokine release syndrome (CRS).

The key features of study design are listed below.

1. Uncontrolled
2. Blinding: open-label
3. Randomized: no
4. Duration of treatment: single infusion within day
5. Titration: none
6. Single center, Taiwan

ELIGIBILITY:
Inclusion Criteria for Enrollment:

A subject may participate in the study if all the following criteria is met:

* Patients with CD19+ malignancies that are refractory to or relapsed after current standard treatment (including allogeneic or autologous HSCT) and not suitable for other treatment options, such as second-time HSCT. CD19+ malignancies include:

  1. Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia (ALL):

     1. Refractory ALL is defined as failure to achieve CR at the end of induction.
     2. Relapsed ALL is defined as reappearance of blasts in the blood or bone marrow (≥ 5%) or in any extramedullary site after a CR.
  2. Relapsed/Refractory B-cell originated Non-Hodgkin Lymphoma (NHL) including 1) de-novo diffuse large B-cell lymphoma or primary mediastinal large B-cell lymphoma, 2) large-B cell lymphoma transformed from indolent lymphomas, 3) follicular lymphoma of all grades, 4) mantle cell lymphoma, and 5) CD20(+) high-grade B-cell lymphomas. Refractory disease for lymphoma is defined as:

     1. Progressive disease or stable disease lasting < 6 months, as best response to most recent chemotherapy regimen; or disease progression or recurrence < 12 months after prior autologous HSCT.
     2. Prior therapy must have included an anti-CD20 monoclonal antibody-containing regimen and an anthracycline-containing chemotherapy regimen
     3. For patients with transformed follicular lymphoma (TFL), prior chemotherapy for follicular lymphoma and subsequent refractory disease after transformation to DLBCL.
     4. At least one measurable lesion, demonstrating that the nodal lesion is ≥ 1.5 cm in the longest diameter or the extranodal lesion is ≥ 1.0 cm in the longest diameter, according to the Lugano Classification (2014).
* Patients must have received at least 2 prior lines of therapy. HSCT (allogeneic or autologous) can be accounted as one of the prior line therapy, and the subjects must have been at least 3 months from prior HSCT.
* Karnofsky Performance Scale ≥ 60
* Patient able to provide written informed consent for participating in the study
* Age ≥ 20 years and ≤ 75 years old at the time of providing informed consent
* Patients shall be at least 3 weeks from the last cytotoxic chemotherapy before apheresis. Short-acting targeted therapies (e.g., tyrosine kinase inhibitors) must be stopped > 72 hours before apheresis.
* Monoclonal antibody use including Anti-CD20 therapy has been discontinued at least 4 weeks before leukapheresis and CAR-T cells infusion except for systemic inhibitory/stimulatory immune checkpoint therapy. Immune checkpoint therapy has been discontinued at least 3 half-lives before leukapheresis (e.g. ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc.).
* Absolute lymphocyte count (ALC) ≥ 1.0x109/L and absolute number of CD3+ T cells (ATC) ≥ 0.3x109/L, absolute neutrophil count (ANC) ≥ 1.0 x109/L for lymphoma and ANC ≥ 0.5 x109/L for ALL, platelets ≥ 50.0 x109/L, hemoglobin ≥ 80.0 g/L within 7 days before apheresis.
* Adequate organ function demonstrated by the following:

  1. Renal: serum creatinine <2 x upper limit of normal (ULN)
  2. Hepatic: ALT/AST ≤ 2.5 x ULN or ≤ 5 x ULN if documented liver metastases, total bilirubin ≤ 1.5 mg/dL, except in subjects with Gilbert's Syndrome in whom total bilirubin must be ≤ 3.0 mg/dL.
  3. Cardiac: no clinically significant ECG findings, hemodynamically stable and LVEF ≥ 45% confirmed by echocardiogram
  4. Pulmonary: baseline oxygen saturation > 90% on room air
* 10. Not receiving anti-thymocyte globulin (ATG), alemtuzumab, or other T-cell immunosuppressive antibodies, donor-lymphocyte infusion or T-cell infusion for the past 3 weeks before apheresis;
* Negative serology for Anti-HTLV-I / HTLV-II (DHTLV I/II)

Exclusion Criteria for Enrollment

A subject who met any of the following criteria is not eligible to enter the study:

* Received previous treatment with anti-CD19 therapy;
* Is with a history of CNS malignancy and/or active CNS diseases;
* Has previous or concurrent malignancies other than CD19+ malignancies;
* Has active neurological, autoimmune, or inflammatory disorders;
* Has clinically significant cardiac diseases, or cardiac arrhythmia not controlled with medical treatment;
* Has cardiac involvement with lymphoma;
* Has any active infections, conditions, and diseases that may interfere with the assessment of safety and efficacy of the study deemed by the investigator or designee;
* Received live vaccine within 6 weeks of the screening
* Received radiation therapy within 2 weeks of the planned CAR-T cells infusion;
* Is with positive serology for HIV;
* Is with positive hepatitis B or hepatitis C infection, defined as positive HBs Ag or positive Anti-HCV Ab;
* Active graft versus host disease (GVHD) ≥ grade 2 using the CIBMTR Acute GVHD Grading System or requiring systemic steroid therapy greater than physiologic dosing; Note: Overall grading of GVHD is based on the criteria published by Przepiorka et al., Bone Marrow Transplant 1995; 15(6):825-8, see the GVHD Grading and Staging table at CIBMTR Forms Instruction Manual (Last updated: 2020/03/10), page 301-303 (Available at https://www.cibmtr.org/manuals/fim, accessed on 08 Apr 2020).
* Use of investigational medicinal product within 30 days before the screening;
* Positive beta HCG in female of child-bearing potential (defined as not post-menopausal for 12 months) or history of previous surgical sterilization or lactating females.
* Patients with known allergy to mouse products or cetuximab.

Inclusion Criteria for Lymphodepletion and T-Cell Infusion:

* Prior to Lymphodepletion (LD):

  1. Patients must have no evidence of clinically significant infection;
  2. No acute neurological toxicity >grade 1 (with the exception of peripheral sensory neuropathy) prior to conditioning chemotherapy;
  3. No clinically significant cardiac dysfunction;
  4. Serum creatinine < 2x ULN;
  5. No evidence of grade ≥2 acute GVHD;
  6. Pulmonary: oxygen saturation > 90% on room air;
  7. Adequacy of T cells apheresis products to manufacture CAR-T product.
* Prior to CAR-T cells infusion:

  1. Patients shall be at least 4 weeks from the last cytotoxic chemotherapy (excluding the study mandated lymphodepleting chemotherapy) before infusion. Short-acting targeted therapies (e.g., tyrosine kinase inhibitors) must be stopped > 72 hours before infusion.
  2. At least 4 weeks from anti-thymocyte globulin (ATG), alemtuzumab, or other T-cell immunosuppressive antibodies, donor-lymphocyte infusion or T-cell infusion;
  3. Steroids, if given as GVHD therapy, must be stopped >72 hours prior to infusion. However, the following physiological replacement doses of steroids are allowed: < 6-12 mg/m2/day hydrocortisone or equivalent.
  4. Non-hematologic toxicity grade ≥2 (CTCAE version 5) related to the lymphodepleting chemotherapy until the toxicity has resolved to grade ≤1 and the subject is afebrile;
  5. No grade >2 neurologic, pulmonary, cardiac, gastrointestinal, renal, or hepatic (excluding albumin) toxicity;
  6. Adequacy of the CAR-T cells for infusion.

Exclusion Criteria For Lymphodepletion and T-Cell Infusion:

A subject who meets any of the following criteria should not undergo LD or infusion of CAR-T cells.

* New onset of cardiac arrhythmia not uncontrolled with medications;
* Hypotension warrants the use of vasopressor;
* Active infections within 1 week prior to CAR-T infusion that necessitate the use of oral or intravenous anti-infective treatments; subjects with ongoing use of prophylactic antibiotics, antifungals, or antivirals are eligible as long as there is no evidence of active infection.
* Presence of CNS or neurological abnormalities;
* Received HSCT after screening or planned to receive HSCT during the study period;
* Any conditions not suitable for the CAR-T cells infusion in the PI or designee's judgement.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Maximun Tolerated Dose (MTD) of the RPM CD19- mbIL15-CAR-T | within 4 weeks after infusion
  MTD is the highest dose at which no more than 1 of 6 patients experiences a dose limiting toxicity.

SECONDARY OUTCOMES:
Feasibility of the product manufacturing process | day 0 to month 12
  Percentage of subjects for whom the desired dose of RPM CD19 mbIL15 CAR-T cells can be successfully manufactured.
Adverse events related to treatment | day 0 to month 12
  The incidence and severity of AE of Cytokine Release Syndrome and neurotoxicity.
Persistence of infused T cells | day 0 to month 12
  Duration of CAR-T cell persistence by vector copy number (VCN).
Safety Switch Function | day 0 to month 12
  Measure the decrease of RPM CD19 mbIL15-CAR-T cells after cetuximab administration.
Immunogenicity | day 0 to month 12
  Immnuogenicity (humoral) defined as the percent of subjects that develop anti-drug antibodies.
Cytokine Profile | day 0 to month 12
  levels of cytokine in serum, including IL-6, IL-10, IFN-γ, TNFα concentration (pg/mL), measured by Elisa.
Homing ability of the infused T-cells | day 0 to month 12
  Percent of subjects with measurable RPM CD19 mbIL15 CAR-T cells in bone marrow.
Disease response after T cell infusion | day 0 to month 12
  Objective response rate (ORR), complete response (CR), Complete response with incomplete blood count recovery (CRi), partial response (PR)
Progression-Free Survival | day 0 to month 12
  Measured from infusion of RPM CD19 mbIL15 CAR-T cells until the documentation of disease progression or death due to any cause, whichever occurs first.
Overall Survival | day 0 to month 12
  Overall survival will be determined as time fro the start of RPM CD19-mbIL15-CAR-T cells infusion until death due to any cause.
Emergence of CD19neg malignant B cells | day 0 to month 12
  CD19 expression of tumor tissue when tumor relapse and progress.

CONTACTS AND LOCATIONS:
Overall Officials: Shangru Wu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No